CLINICAL TRIAL: NCT00114114
Title: Dose-Response of Gonadal Steroids and Bone Turnover in Older Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Solvay Pharmaceuticals (Industry); AstraZeneca (Industry); AbbVie (Industry)
Responsible Party: Principal Investigator, Benjamin Leder, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2003-P-001868; R01AG030545 (NIH)
Record Dates: First submitted 2005-06-13; First posted 2005-06-14 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Healthy Volunteers
Keywords: Testosterone; Bone turnover; Aging; Body composition; Hypogonadism; Sexual function
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone; Goserelin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1: 0 g/day (Experimental): Zoladex plus Placebo Testosterone (T) gel
  Interventions: Drug: Testosterone; Drug: Goserelin acetate
- Group 2: 1.25 g/day (Experimental): Zoladex plus 1.25 g/day T gel
  Interventions: Drug: Testosterone; Drug: Goserelin acetate
- Group 3: 2.5 g/day (Experimental): Zoladex plus 2.5 g/day T gel
  Interventions: Drug: Testosterone; Drug: Goserelin acetate
- Group 4: 5 g/day (Experimental): Zoladex plus 5 g/day T gel
  Interventions: Drug: Testosterone; Drug: Goserelin acetate
- Group 5: 10* g/day (Experimental): Zoladex plus 10* g/day T gel. *Note that the 10 g/day dose was reduced to 7.5 g/day part-way through the trial
  Interventions: Drug: Testosterone; Drug: Goserelin acetate
- Group 6: Placebo/Placebo (PBO/PBO) (Experimental): Placebo Zoladex plus Placebo T gel (controls)
  Interventions: Drug: Testosterone; Drug: Goserelin acetate

INTERVENTIONS:
Drug: Testosterone — Androgel placebo or 1.25, 2.5, 5. or 10* gms topically each day
  Other Names: Androgel
Drug: Goserelin acetate — 3.6 gms sc every 4 weeks
  Other Names: Zoladex

SUMMARY:
The purpose of this study is to determine the levels of testosterone and/or estradiol at which changes in bone turnover, body composition, strength, sexual function etc. begin to occur in older men. This information may help determine when to intervene with hormone replacement therapy in aging men.

DETAILED DESCRIPTION:
In this protocol, men age 60-75 will be randomized to one of 6 groups. Groups 1-5 will receive goserelin acetate (Zoladex) plus 0 (placebo gel), 1.25, 2.5, 5, or 10* g/day of testosterone gel (Androgel). Group 6 will receive placebos for both goserelin acetate and testosterone gel. (*Note that the 10 g/day dose was reduced to 7.5 g/day part-way through the trial due to reports of possible increased risk of cardiovascular events with testosterone administration).

Subjects will be blinded with respect to group assignment. Dietary calcium intake will be assessed by a research dietitian and adjustments made through diet or supplements so that calcium intake is between 1000 and 1200 mg/day.

Subjects will be seen on the Clinical Research Center at 4 week intervals for 16 weeks (0, 4, 8, 12, and 16 weeks). At each visit, compliance with Androgel will be assessed by reviewing a medication diary. A standardized series of questions will be posed to each subject to assess potential side effects of the study drugs. Subjects receiving Androgel' will be given a new 4 week supply of medication (except at week 16). A fasting blood and second voided urine sample will be collected. After the blood and urine samples have been obtained, subjects will be given their goserelin injection. The blood and urine tests listed below as well as anthropometric measures, and questionnaires will be performed at each visit. Dual-energy x-ray absorptiometry (DXA), quantitate computed tomography (QCT) scans, and strength assessments will be performed at 0 and 16 weeks only. Subjects who discontinue participation at or after week 8 will be asked if they are willing to have an early discontinuation visit in which all procedures normally done at week 16 will be performed.

The following measures will be assessed:

* Routine chemistries and prostate specific antigen, PSA (for safety assessment)
* Bone turnover using blood and urine tests
* Hormones
* Lipids
* Body composition
* Strength
* Sexual desire and erectile function
* Bone mineral density and bone microarchitecture

ELIGIBILITY:
Inclusion Criteria:

* Healthy men age 60 to 75

Exclusion Criteria:

* History of significant cardiac, renal, pulmonary, hepatic, benign prostatic hyperplasia, or malignant disease, current alcohol or illicit drug abuse, or major psychiatric disorders.
* Current diagnoses of disorders known to affect bone metabolism including hyperthyroidism, hyperparathyroidism, osteomalacia, or Paget's disease.
* Current use of medications known to affect bone metabolism including estrogens, androgens, anti-estrogens, bisphosphonates, calcitonin, fluoride, oral or inhaled glucocorticoids, suppressive doses of thyroxine, lithium, pharmacological doses of vitamin D (greater than 2000 IU/day), or anti-convulsants.
* Cognitive or intellectual impairment that precludes complete understanding of the study protocol.
* History of deep vein thrombosis, pulmonary embolism, or clotting disorders.
* Serum 25-hydroxyvitamin D < 15 ng/mL
* Serum parathyroid hormone (PTH) < 10 or > 65 pg/mL
* Serum thyroid stimulating hormone (TSH) < 0.5 or > 5.0 U/L
* Serum calcium > 10.6 mg/dL
* Serum creatinine > 2 mg/dL
* Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 2x the upper limit of normal
* Serum bilirubin > 2 mg/dL
* Serum alkaline phosphatase > 150 U/L
* Plasma hemoglobin < 11 gm/dL
* Hematocrit > 50
* Fracture within the last 6 months.
* Serum testosterone level < 270 or > 1070 ng/dL
* Serum prostate specific antigen (PSA) level > 4 ug/L.
* International Prostate Symptom Score (IPSS) > 19
* Systolic blood pressure > 160 or diastolic blood pressure > 95
* Framingham risk score greater than or equal to 20
* Difficulty walking 2 blocks

Ages: 60 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2004-09; Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ben Z Leder, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Finkelstein JS, Lee H, Burnett-Bowie SM, Darakananda K, Gentile EC, Goldstein DW, Prizand SH, Krivicich LM, Taylor AP, Wulczyn KE, Leder BZ, Yu EW. Dose-Response Relationships Between Gonadal Steroids and Bone, Body Composition, and Sexual Function in Aging Men. J Clin Endocrinol Metab. 2020 Aug 1;105(8):2779-88. doi: 10.1210/clinem/dgaa318. PMID 32480409
- [Derived] Bachmann KN, Huang S, Lee H, Dichtel LE, Gupta DK, Burnett JC Jr, Miller KK, Wang TJ, Finkelstein JS. Effect of Testosterone on Natriuretic Peptide Levels. J Am Coll Cardiol. 2019 Mar 26;73(11):1288-1296. doi: 10.1016/j.jacc.2018.12.062. PMID 30898204
- [Derived] Finkelstein JS, Lee H, Leder BZ, Burnett-Bowie SA, Goldstein DW, Hahn CW, Hirsch SC, Linker A, Perros N, Servais AB, Taylor AP, Webb ML, Youngner JM, Yu EW. Gonadal steroid-dependent effects on bone turnover and bone mineral density in men. J Clin Invest. 2016 Mar 1;126(3):1114-25. doi: 10.1172/JCI84137. Epub 2016 Feb 22. PMID 26901812
- [Derived] Finkelstein JS, Lee H, Burnett-Bowie SA, Pallais JC, Yu EW, Borges LF, Jones BF, Barry CV, Wulczyn KE, Thomas BJ, Leder BZ. Gonadal steroids and body composition, strength, and sexual function in men. N Engl J Med. 2013 Sep 12;369(11):1011-22. doi: 10.1056/NEJMoa1206168. PMID 24024838

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: 0 Grams/Day: Zoladex plus Placebo T gel
- Group 5: 10* g/Day: Zoladex plus 10 g/day T gel; *Note that the 10 g/day dose was reduced to 7.5 g/day part-way through the trial
- Group 6: PBO/PBO: Placebo Zoladex plus Placebo T gel
Period: Overall Study
Arm/Group | Group 1: 0 Grams/Day | Group 2: 1.25 g/Day | Group 3: 2.5 g/Day | Group 4: 5 g/Day | Group 5: 10* g/Day | Group 6: PBO/PBO
Started | 26 | 25 | 31 | 35 | 29 | 31
Completed | 21 | 24 | 30 | 31 | 27 | 30
Not Completed | 5 | 1 | 1 | 4 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group 1: 0 g/Day: Zoladex plus Placebo T gel
- Group 5: 10* g/Day: Zoladex plus 10* g/day T gel; *Note that the 10 g/day dose was reduced to 7.5 g/day part-way through the trial
- Total: Total of all reporting groups
Arm/Group | Group 1: 0 g/Day | Group 2: 1.25 g/Day | Group 3: 2.5 g/Day | Group 4: 5 g/Day | Group 5: 10* g/Day | Group 6: PBO/PBO | Total
Number analyzed (Participants) | 26 | 25 | 31 | 35 | 29 | 31 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (5) | 64 (3) | 64 (4) | 65 (4) | 65 (3) | 65 (4) | 65 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 26 | 25 | 31 | 35 | 29 | 31 | 177
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 35 | 0 | 0 | 39
  Not Hispanic or Latino | 25 | 23 | 29 | 0 | 28 | 30 | 135
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 0 | 4 | 1 | 0 | 8
  White | 26 | 22 | 29 | 31 | 28 | 29 | 165
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 25 | 31 | 35 | 29 | 31 | 177
Height [Mean (Standard Deviation); unit: cm] | 175.2 (5.7) | 175.1 (8.7) | 176.5 (7.9) | 177.5 (7.6) | 175.4 (5.0) | 176.7 (6.5) | 176.2 (7.0)
Weight [Mean (Standard Deviation); unit: kg] | 86.2 (14.1) | 83.9 (15.0) | 82.0 (14.2) | 85.7 (15.1) | 86.8 (12.2) | 83.9 (13.0) | 84.8 (13.9)
Body-mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.0 (3.9) | 27.3 (4.3) | 26.3 (4.3) | 27.1 (4.2) | 28.2 (3.5) | 26.9 (4.2) | 27.3 (4.1)
Testosterone [Mean (Standard Deviation); unit: ng/dL] | 496 (176) | 485 (117) | 491 (142) | 483 (165) | 484 (148) | 505 (155) | 490 (150)
Estradiol [Mean (Standard Deviation); unit: pg/mL] | 27 (7) | 26 (11) | 25 (8) | 30 (11) | 26 (6) | 28 (7) | 27 (9)
Total-body Lean Mass [Mean (Standard Deviation); unit: g] | 56177 (6417) | 55553 (8218) | 55428 (8054) | 55653 (9206) | 56081 (6116) | 55867 (6637) | 55784 (7444)
Total body fat mass [Mean (Standard Deviation); unit: g] | 22773 (8693) | 20827 (7208) | 19396 (7567) | 23062 (11123) | 22803 (7459) | 19931 (7574) | 21471 (8564)
Thigh-muscle area [Mean (Standard Deviation); unit: mm^2] | 15272 (2026) | 16006 (2515) | 15281 (2645) | 15367 (2820) | 15771 (2145) | 15572 (2157) | 15531 (2424)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Bone Turnover Marker (Serum C-telopeptide, CTX)
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Error); unit: percentage change
Groups:
- Group 6: Placebo/Placebo (PBO/PBO): Placebo Zoladex plus Placebo T gel
Arm/Group | Group 1: 0 g/Day | Group 2: 1.25 g/Day | Group 3: 2.5 g/Day | Group 4: 5 g/Day | Group 5: 10* g/Day | Group 6: Placebo/Placebo (PBO/PBO)
Number analyzed (Participants) | 21 | 24 | 30 | 31 | 27 | 30
percentage change | 103 (12) | 41 (6) | 29 (6) | 15 (7) | 4 (5) | 11 (6)

2. Secondary Outcome: Percentage Change in Body Composition: Fat Mass
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Error); unit: Percentage change
Arm/Group | Group 1: 0 g/Day | Group 2: 1.25 g/Day | Group 3: 2.5 g/Day | Group 4: 5 g/Day | Group 5: 10* g/Day | Group 6: PBO/PBO
Number analyzed (Participants) | 21 | 24 | 30 | 31 | 27 | 30
Percentage change | 9.8 (2.4) | 5.7 (1.1) | 1.9 (1.5) | 0.4 (1.3) | -1.6 (1.6) | 2.3 (1.9)

3. Secondary Outcome: Percentage Change in Thigh Muscle Area
Description: Assessed by quantitative computed tomography (QCT)
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Group 1: 0 g/Day | Group 2: 1.25 g/Day | Group 3: 2.5 g/Day | Group 4: 5 g/Day | Group 5: 10* g/Day | Group 6: PBO/PBO
Number analyzed (Participants) | 21 | 24 | 30 | 31 | 27 | 30
percentage change | -1.5 (1.1) | -1.6 (0.9) | -0.4 (0.5) | -0.5 (0.7) | 0.5 (0.7) | -0.9 (0.6)

4. Secondary Outcome: Change in Erectile Function Symptoms
Description: Based on International Index of Erectile Function (IIEF) scale, question #15, which asked subjects to rate their confidence that they could achieve and maintain an erection. Scores range from 1 to 5, with higher scores being better.
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Group 1: 0 g/Day | Group 2: 1.25 g/Day | Group 3: 2.5 g/Day | Group 4: 5 g/Day | Group 5: 10* g/Day | Group 6: PBO/PBO
Number analyzed (Participants) | 21 | 24 | 30 | 31 | 27 | 30
units on a scale | -1.4 (0.2) | -0.5 (0.2) | -0.2 (0.2) | -0.1 (0.2) | 0.2 (0.2) | -0.3 (0.2)

5. Secondary Outcome: Change in Libido / Sexual Desire
Description: Change in libido from baseline (scale ranges from -2 to +2), with -2 being much less, -1 somewhat less, 0 same, +1 somewhat more, +2 much more
Time Frame: 16 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Group 1: 0 g/Day | Group 2: 1.25 g/Day | Group 3: 2.5 g/Day | Group 4: 5 g/Day | Group 5: 10* g/Day | Group 6: PBO/PBO
Number analyzed (Participants) | 21 | 24 | 30 | 31 | 27 | 30
units on a scale | -1.6 (0.2) | -0.6 (0.2) | -0.6 (0.2) | -0.2 (0.2) | 0 (0.1) | -0.3 (0.1)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Group 1: 0 g/Day | Group 2: 1.25 g/Day | Group 3: 2.5 g/Day | Group 4: 5 g/Day | Group 5: 10* g/Day | Group 6: PBO/PBO
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25 | 0/31 | 0/35 | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25 | 0/31 | 0/35 | 0/29 | 0/31
Other Adverse Events (participants affected / at risk) | 3/26 | 0/25 | 0/31 | 1/35 | 2/29 | 0/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: 0 g/Day (N=26) | Group 2: 1.25 g/Day (N=25) | Group 3: 2.5 g/Day (N=31) | Group 4: 5 g/Day (N=35) | Group 5: 10* g/Day (N=29) | Group 6: PBO/PBO (N=31)
Increased Prostate Specific Antigen (PSA) (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) — PSA >=4 ng/mL or whose PSA increased by >= 1 ng/mL

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT00114114/Prot_SAP_000.pdf